CLINICAL TRIAL: NCT00466622
Title: Uterine Artery Blood Flow in Pregnant Women With Polycystic Ovary Syndrome(PCOS)Treated With Metformin - a Substudy to The PregMet Study
Brief Title: Uterine Artery Blood Flow in Pregnant Women With PCOS Treated With Metformin
Acronym: FlowMet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2004-000792-33
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; pregnancy; metformin; blood flow; Pulsatility index
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Metformin 1000mg x 2 daily. Orally. From Weifa
  Interventions: Drug: Metformin
- 2 (Placebo Comparator): Placebo 2 tablets x 2 daily. Orally From Weifa
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 1000 mg x 2 daily. Orally. First tablet taken after the first Doppler examination and 3 hours before the next Doppler examination.
  Other Names: metformin 500mg tablets from Weifa
  Arms: 1
Drug: Placebo — Placebo 2 tablets x 2 daily. Orally from Weifa
  Other Names: Placebo tablets from Weifa
  Arms: 2

SUMMARY:
FlowMet study is a "sub-study" of the PregMet study (registered in 2005).

The aim of the FlowMet study is to register the possible effect of metformin on the blood flow of the uterine artery in pregnant PCOS women. The participants will be examined with ultrasound Doppler in gestational week 10-13:

1. before and 3h after the first tablet intake of metformin/placebo
2. and 10-14 days after inclusion in the trial
3. blood flow in the umbilical artery and fetal cerebral artery in gestational week 24.

ELIGIBILITY:
Inclusion Criteria:

* Same as in the PregMet study. As this study is a sub-study/extended study of the PregMet study, ONLY those included in the PregMet study (NCT00159536) can participate.

Exclusion Criteria:

* Same as in the PregMet study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pulsatility index of the uterine artery | up to delivery
  3 hrs before and after drug intake, 2 weeks after inclusion, and during medication

SECONDARY OUTCOMES:
Blood flow in the umbilical artery and fetal cerebral artery | 24 weeks gestational

CONTACTS AND LOCATIONS:
Overall Officials: Eszter Vanky, MD, Phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Dept. of Obstetrics and Gynecology, National Center for fetal Medicine, University Hospital of Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Stridsklev S, Carlsen SM, Salvesen O, Clemens I, Vanky E. Midpregnancy Doppler ultrasound of the uterine artery in metformin- versus placebo-treated PCOS women: a randomized trial. J Clin Endocrinol Metab. 2014 Mar;99(3):972-7. doi: 10.1210/jc.2013-3227. Epub 2014 Jan 1. PMID 24423336
- [Derived] Stridsklev S, Salvesen O, Salvesen KA, Carlsen SM, Vanky E. Uterine Artery Doppler in Pregnancy: Women with PCOS Compared to Healthy Controls. Int J Endocrinol. 2018 Aug 16;2018:2604064. doi: 10.1155/2018/2604064. eCollection 2018. PMID 30186323